CLINICAL TRIAL: NCT01040754
Title: An fMRI Study of Expectancy on Acupuncture Treatment Outcomes in Knee OA
Brief Title: fMRI Study of Expectancy on Acupuncture Treatment Outcomes in Knee OA
Acronym: KOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Randy L. Gollub, Clinical Associate at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2009P000096; R01AT005280 (NIH)
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Active Comparator)
  Interventions: Other: Acupuncture
- Waitlist Control (No Intervention)

INTERVENTIONS:
Other: Acupuncture — This study follows a standardized acupuncture protocol for OA knee pain. Approximately 6 acupuncture needles are placed in the skin of the leg for 25 minutes.
  Arms: Acupuncture

SUMMARY:
The results of the proposed experiments will directly inform clinicians who treat patients with osteoarthritis of the knee about how to maximize the benefits of acupuncture treatments. And because the experiments specifically asks the question of what is the relation between a patient's expectation of how a treatment will relieve their pain and the outcome of the treatment, the results will potentially inform care givers about all treatments for osteoarthritis and other chronic pain disorders. We hypothesize that acupuncture treatment will produce clinically significant analgesia as indicated by lowered sensory ratings of noxious stimuli and endogenous knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers 40-70 years of age.
* Meet the Classification Criteria of the American College of Rheumatology for osteoarthritis of the right and/or left knee for at least the past 3 months, as determined by the referring physician.
* Radiographic evidence of Grade 2 or 3 knee OA using the Kellgren-Lawrence Scale.
* Ability to read and understand English; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Any interventional procedure for knee pain, including corticosteroid injections (within 2 months) to the knee.
* Prior acupuncture treatment for any condition. Because we are using a placebo needle as a control, acupuncture-naive patients are necessary to maximize the benefits of blinding and to control expectancy.
* The intent to undergo surgery during the time of involvement in the study.
* Presence of any illness or medication use that is judged to interfere with the trial. For example: skin irritations around the knee such as psoriasis; bleeding disorders or anticoagulant use that would be contraindications for acupuncture; diabetes due to the increased possibility of sensitivity to heat pain; and use of opiate medications and other substances of abuse that may influence the patient's experience of analgesia. (Due to the potential risk that prescription or non-prescription medication use can confound our results, we may perform a urine toxicology screen to verify patient's medication status during Session 1.)
* Knee pain due to other causes, such as inflammation or malignancy, other pain disorders that may refer pain to the leg, OA of ipsilateral hip, diagnosis of rheumatoid arthritis (RA).
* Non-ambulatory status.
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome. For example: asthma or claustrophobia.
* Presence of any contraindications to fMRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy.
* Instability of pain rating within Session 1 or Session 2 of Experiment One or Visit 1 of Experiment Two.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2009-06; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The difference (pre- minus post-treatment) in subjective pain rating and fMRI BOLD response to calibrated experimental noxious stimuli (noxious heat and pressure) used as a proxy for endogenous knee pain. | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Randy L Gollub, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided